CLINICAL TRIAL: NCT03243981
Title: Augmentation of Skin Aging Reversal By Broadband Light With Skin Tightening Properties Via Gene Expression Analysis
Brief Title: Infrared and Broadband Light for Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Sciton (Industry)
Responsible Party: Principal Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 37776
Record Dates: First submitted 2017-07-11; First posted 2017-08-09 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Application of Skintyte and/or broadband light to skin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Open label study-- single arm (Experimental): All patients will receive Skintyte treatment as well as Skintyte plus broadband light
  Interventions: Device: Sciton SkinTyte (800-1800 nm) with Broadband Light Technology

INTERVENTIONS:
Device: Sciton SkinTyte (800-1800 nm) with Broadband Light Technology — This device has been used in the clinical setting to reduce cheek and submental laxity. SkinTyte delivers sequentially pulsed light (800-1200 nm, with a filter enabling focus on 590 nm) and broadband light (which can be turned on or off).

SUMMARY:
In this exploratory study, we hope to learn if treatment of broadband light with infrared light can alter the molecular pathways associated with aging. Secondary exploratory objective is to see if there are any visible effects of this light treatment on human skin.

DETAILED DESCRIPTION:
Studies in model organisms suggest that aged cells can be functionally rejuvenated, but whether this concept applies to human skin is unclear. Recently, we applied 3'-end sequencing for expression quantification ("3-seq") to discover the gene expression program associated with human photoaging and intrinsic skin aging (collectively termed "skin aging"), and the impact of broadband light (BBL) treatment. We found significant changes in 2,265 coding and noncoding RNAs, of which 1,293 that became "rejuvenated" after BBL treatment, whereby they became more similar to their expression level in youthful skin. Rejuvenated genes (RGs) included several known key regulators of organismal longevity and their proximal long noncoding RNAs. Hence, BBL treatment can restore gene expression pattern of photo-aged and intrinsically aged human skin to resemble young skin.

However, the duration of these effects and the potential to augment these effects through increases in particular wavelengths of light have not been explored. The Sciton SkinTyte (800-1800nm) is the ideal technology to examine these questions, since this device has been used in the clinical setting to reduce cheek and submental laxity (Gold, 2010). It incorporates the broadband light technology with an emphasis on 590 nm filter to achieve these clinical results.

This study will be conducted in accord with Declaration of Helsinki principles. After Institutional Review Board approval and informed consent is obtained, six female participants over the age of 55 years will undergo BBLST treatments to the left forearm. Inclusion criteria included Fitzpatrick skin type II or III, and a global assessment of forearm skin aging consistent with moderate or severe forearm skin aging (modified validated instrument from McKenzie et al., 2011) for treated participants. Treatments will be performed on the Sciton Joule Platform using BBL in Skintyte mode with 590ST filter. On a separate part of the arm that is clearly marked, Skintyte alone will be applied. Untreated areas will also be marked. All markings will be photographed. The same investigator will perform the treatments at 4-week intervals for a total of 3 treatments. At each treatment session, two or more passes were performed. Four weeks after the third BBL treatment, 4 mm skin biopsies will performed by Keys punch technique from the BBLST treated, ST treated and adjacent untreated skin. These specimens will be bisected and placed into either RNAlater (Ambion Cat# AM7022) or formalin solution for with H&E, von Giesen or PAS staining.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female 2. Age 55 years or older (total 6) 3. Fitzpatrick skin type 2-3 4. Photo-aging at least moderate on the extensor forearms

Exclusion Criteria:

* 1. Unable to understand and sign informed consent form 2. Unable to comply with study procedures 3. Pregnant or lactating 4. Prior treatment to forearms including topical retinoid, laser treatment, photodynamic treatment, prescription topical agents x 1 month 5. Active skin conditions that precluding treatment including zoster, blistering skin disease, psoriasis, atopic dermatitis, abnormal scarring, skin cancer in the area of study treatment 6. Currently on hormone based therapy (both systemic and topical)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Skintyte: All patients will receive Skintyte treatment as well as Skintyte plus broadband light using the Sciton SkinTyte device.
Period: Overall Study
Arm/Group | Skintyte
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Skintyte
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Genes With Significant Change in Gene Transcription
Description: The endpoint consisted of clinical inspection of biopsies of untreated skin and skin after three treatments. Genes were considered altered if a statistically significant change in transcription of an individual gene was observed between the treated and untreated skin (significance was set at p<0.01, adjusted for false discovery rate). The values in the table represent the total number of recorded genes with significant change.
Time Frame: 16 weeks
Measure: Number; unit: genes
Groups:
- BBL + SPL590 vs Untreated: Biopsies were collected from the BBL + SPL590-treated arm (proximal forearm) and the untreated arm (mid-forearm)
  BBL = broadband light; SPL = sequentially pulsed light
- SPL800 (SkinTite 2) vs Untreated: Biopsies were collected fro the SPL800-treated arm (distal forearm) vs untreated arm (mid-forearm)
  SPL800 = SkinTite 2
Arm/Group | BBL + SPL590 vs Untreated | SPL800 (SkinTite 2) vs Untreated
Number analyzed (Participants) | 5 | 5
genes | 188 | 45

2. Secondary Outcome: Change From Baseline in Fine Wrinkling Score as a Measure of Skin Rejuvenation
Description: Wrinkling was assessed on a 10 point Likert scale (range 1-10); higher scores correspond to more wrinkling.
Time Frame: Baseline, day 84
Population: Participants that had assessments at baseline and day 84 are included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BBL + SPL590: Treatment on proximal forearm
- SPL800: Treatment on distal forearm
Arm/Group | BBL + SPL590 | SPL800
Number analyzed (Participants) | 4 | 4
score on a scale
  Baseline | 7.8 (1.89) | 7.5 (3.70)
  Day 84 | 5.0 (3.46) | 5.3 (3.20)

3. Secondary Outcome: Change From Baseline in Coarse Wrinkling Score as a Measure of Skin Rejuvenation
Description: Wrinkling was assessed on a 10 point Likert scale (range 1-10); higher scores correspond to more wrinkling.
Time Frame: Baseline, day 84
Population: Participants that had assessments at baseline and day 84 are included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BBL + SPL590 | SPL800
Number analyzed (Participants) | 4 | 4
score on a scale
  Baseline | 5.0 (3.65) | 6.0 (1.83)
  Day 84 | 2.3 (2.63) | 2.5 (1.73)

4. Secondary Outcome: Change From Baseline in Sagging Score as a Measure of Skin Rejuvenation
Description: Sagging was assessed on a 10 point Likert scale (range 1-10); higher scores correspond to more sagging.
Time Frame: Baseline, day 84
Population: Participants that had assessments at baseline and day 84 are included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BBL + SPL590 | SPL800
Number analyzed (Participants) | 4 | 4
score on a scale
  Baseline | 7.0 (1.63) | 7.5 (1.91)
  Day 84 | 3.5 (1.73) | 4.3 (2.06)

5. Secondary Outcome: Change From Baseline in Physician Global Assessment as a Measure of Skin Rejuvenation
Description: Physician global assessment was assessed on a 10 point Likert scale (range 1-10); higher scores correspond to more severe skin aging.
Time Frame: Baseline, day 84
Population: Participants that had assessments at baseline and day 84 are included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BBL + SPL590 | SPL800
Number analyzed (Participants) | 4 | 4
score on a scale
  Baseline | 8.3 (0.96) | 8.3 (1.50)
  Day 84 | 5.5 (2.08) | 6.0 (1.83)

6. Secondary Outcome: Change From Baseline in Cutometry as a Measure of Skin Rejuvenation
Description: Elasticity of skin assessment with cutometric probe.
Time Frame: Baseline, day 84
Population: Data were not collected for this outcome
Arm/Group | BBL + SPL590 | SPL800
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Transepidermal Water Loss as a Measure of Skin Rejuvenation
Description: Transepidermal water loss assessment with VapoMeter.
Time Frame: Baseline, day 84
Population: Data were not collected for this outcome
Arm/Group | BBL + SPL590 | SPL800
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Groups:
- Untreated: Untreated area on mid-forearm
Arm/Group | BBL + SPL590 | SPL800 | Untreated
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The study did not meet its planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03243981/Prot_SAP_000.pdf